CLINICAL TRIAL: NCT05235373
Title: Prognostic Significance of COVID-19 MSCT Chest Findings on Short Term Disease Progression
Acronym: MSCT
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, AMIRA HUSSEIN ALLAM, assistant professor of chest diseases and tuberculosis, Benha University
Other Study IDs: TEJB-D-22-00019
Record Dates: First submitted 2022-02-08; First posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Infection Viral
Keywords: COVID-19; MSCT; chest
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group A: (mild cases): with no progression of the respiratory symptoms.: multislice CT finding,The CT finding were then compared to the short-term clinical outcome of the patients (1-3weeks), acquired from the hospital patient data archive.
- group B: (moderate cases): who have worsened disease but not requiring ICU admission.: multislice CT finding,The CT finding were then compared to the short-term clinical outcome of the patients (1-3weeks), acquired from the hospital patient data archive.
- Group C: (sever cases): patient who needed ICU admission.: multislice CT finding,The CT finding were then compared to the short-term clinical outcome of the patients (1-3weeks), acquired from the hospital patient data archive.
- Group D: (fatality cases): cases who died with or without ICU admission).: multislice CT finding,The CT finding were then compared to the short-term clinical outcome of the patients (1-3weeks), acquired from the hospital patient data archive.

SUMMARY:
Background: CT has been used on a massive scale to help identify and investigate suspected or confirmed cases of COVID-19 pneumonia. This study aimed to assess the prognostic significance of the chest findings MSCT of Covid-19 patients and to determine if prognosis can rely on the initial CT imaging. Methods: The study design was retrospective cohort study. It was carried out on 300 patients presented to the chest outpatient clinics in Benha university hospitals and Elabbasyia chest hospital with clinical picture suggestive of COVID 19 infection. The CT finding were then compared to the short-term clinical outcome of the patients (1-3weeks), acquired from the hospital patient data archive. According to the progression of the respiratory symptoms (include; dyspnea, respiratory rate and O2 saturation), the short-term clinical outcome of the patients was classified into 4 groups; Group A: (mild cases), Group B: (moderate cases), Group C: (sever cases), and Group D: (fatality cases).

DETAILED DESCRIPTION:
Patients and methods The study design was retrospective cohort study. It was carried out on 300 patients presented to the chest outpatient clinics in Benha university hospitals and Elabbasyia chest hospital with clinical picture suggestive of COVID 19 infection during the period from April 2020 to December 2020.

Inclusion criteria:

• Patients who had positive RT-PCR test for COVID-19 infection and show positive chest CT findings.

Exclusion criteria:

* Patients with negative RT PCR test for COVID 19 infection.
* Patients with positive RT PCR test for COVID 19 and negative chest CT findings.
* Patients with other pre-existing lung pathologies in the chest CT.

Data were collected from patients files included; history including symptoms and co-morbidities , and previously available examination data.

Approval was taken from the ethics committee of researchers of Benha university. An informed consent was taken from all the participants.

The consent contains:

1. Their approval that their studies and clinical data could be used for research purpose.
2. All patients' clinical data is considered confidential.
3. Signatures or fingerprints of the participants were taken. The picture archiving and communication systems (PACS) in both hospitals were revised during the period form the 1st of April 2020 to the 31st of December 2020. The included CT studies were revised first for technical appropriateness, and the studies with technical problems were excluded.

All chest CT examinations were performed using multislice CT equipment (Toshiba Activion 16 and Toshiba Alexion 16). The exams were performed with patients in supine position and breath-hold during full expiration. The scanning range was from the lower neck down to the level of the adrenal glands. The scanning parameters were as follows: helical scanning mode; tube voltage, 120 kV; tube current-time product, 50-350 mAs; pitch, 1.2 and 1.375; matrix, 512 × 512; slice thickness, 5 mm; reconstructed in distribution lung window; reconstructed slice thickness, 1.25 mm. Followed by sagittal and coronal reconstruction.

The technically accepted studies were extracted from the PACS system. They were interpreted by radiologists and pulmonologist (14 and 10 years in chest CT interpretation respectively) in blind manner.

The following CT features were assessed: (peripheral, central, or central and peripheral), number of lobes involved (one, two or three, four or five), shape (patchy, nodular), appearance (ground-glass opacity [GGO], consolidation, or GGO with consolidation), specific signs within the lesions (vascular thickening, crazy paving pattern, air bronchogram sign, halo sign, and fibrosis), size of largest lesion (< 1 cm, 1-3 cm, > 3 cm), and extra-pulmonary manifestations (mediastinal and hilar lymph node enlargement, pleural effusion, pleural thickening). CT severity scoring was calculated for each case (2).

The CT finding were then compared to the short-term clinical outcome of the patients (1-3weeks), acquired from the hospital patient data archive. According to the progression of the respiratory symptoms (dyspnea, respiratory rate and O2 saturation), the short-term clinical outcome of patients was classified into 4 groups, as follows:

1. Group A: (mild cases): with no progression of the respiratory symptoms.
2. Group B: (moderate cases): who have worsened disease but not requiring ICU admission.
3. Group C: (sever cases): patient who needed ICU admission.
4. Group D: (fatality cases): cases who died with or without ICU admission). Statistical Analysis Data were collected, revised, coded and entered to the Statistical Package for Social Science (IBM SPSS) version 20. The qualitative data were presented as number and percentages while quantitative data were presented as mean, standard deviations and ranges when their distribution found parametric. The comparison between two groups with qualitative data were done by using Chi-square test and/or Fisher exact test which was used instead of Chi-square test when the expected count in any cell was found less than 5. The comparison between more than two independent groups with quantitative data and parametric distribution was done by using One Way ANOVA Test. The confidence interval was set to 95% and the margin of error accepted was set to 5%. So, the p-value was considered significant as the following: P> 0.05 = non-significant (NS), P < 0.05 = significant (S), P < 0.001 = highly significant (HS)

ELIGIBILITY:
Inclusion Criteria:• Patients who had positive RT-PCR test for COVID-19 infection and show positive chest CT findings.

-

Exclusion Criteria:• Patients with negative RT PCR test for COVID 19 infection.

* Patients with positive RT PCR test for COVID 19 and negative chest CT findings.
* Patients with other pre-existing lung pathologies in the chest CT.

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: presented to the chest outpatient clinics in Benha university hospitals and Elabbasyia chest hospital with clinical picture suggestive of COVID 19 infection during the period from April 2020 to December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
correlation between initial CT findings with short term clinical outcome | 3 weeks
  The CT finding were then compared to the short-term clinical outcome of the patients (1-3weeks), acquired from the hospital patient data archive; respiratory symptoms (dyspnea, respiratory rate and O2 saturation),

CONTACTS AND LOCATIONS:
Overall Officials: AMIRA HM Allam, MD, Principal Investigator — chest department, Faculty of medicine, Benha University, Egypt
Locations (1):
- Benha University hospital, Banhā, Kalyobia, Egypt

IPD SHARING:
Plan to Share IPD: No